CLINICAL TRIAL: NCT05544370
Title: H2 Physical Education: Promoting Cardiometabolic Health by 2 High Intensity Intervallic Training Protocol, Twice a Week at Physical Education
Acronym: H2PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Noelia González-Gálvez, Principal investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCMurcia-H2PE
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Behavior
Keywords: adolescents; cardiovascular; strength; high intensity interval training; metabolic syndrome; physical activity
MeSH Terms: conditions — Adolescent Behavior; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensive high intensity intervallic training group (Experimental): The intensive high intensity intervallic training group performs 6 sets of 60 seconds of work and 60 seconds of rest. During the first two weeks we work at an intensity of 80-85% of the reserve heart rate during the work phase and 50-55% of the reserve heart rate during the rest time. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 95-95% of the reserve heart rate. The program duration is 8 weeks and the frequency of intervention is 2 sessions per week.
  Interventions: Behavioral: Intensive high intensity intervallic training group
- Extensive high-intensity intervallic training group (Experimental): The extensive high-intensity intervallic training group performs 3 sets of 120 seconds of work and 120 seconds of rest at an intensity of 70-75% of the reserve heart rate during the work phase and an intensity of 50-55% of the reserve heart rate during the rest phase. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 80-85% of the reserve heart rate. The program duration is 8 weeks and the frequency of intervention is 2 sessions per week.
  Interventions: Behavioral: Extensive high-intensity intervallic training
- Control group (No Intervention): The control group will carry out their usual physical education classes which consist of games, jumping, moving, balance and different sports.

INTERVENTIONS:
Behavioral: Intensive high intensity intervallic training group — The intensive high intensity intervallic training group performs 6 sets of 60 seconds of work and 60 seconds of rest. During the first two weeks we work at an intensity of 80-85% of the reserve heart rate during the work phase and 50-55% of the reserve heart rate during the rest time. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 95-95% of the reserve heart rate. The program duration is 8 weeks and the frequency of intervention is 2 sessions per week.
  Arms: Intensive high intensity intervallic training group
Behavioral: Extensive high-intensity intervallic training — The extensive high-intensity intervallic training group performs 3 sets of 120 seconds of work and 120 seconds of rest at an intensity of 70-75% of the reserve heart rate during the work phase and an intensity of 50-55% of the reserve heart rate during the rest phase. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 80-85% of the reserve heart rate. The program duration is 8 weeks and the frequency of intervention is 2 sessions per week.
  Arms: Extensive high-intensity intervallic training group

SUMMARY:
Several risk factors associated with cardiovascular disease could be prevented or treated by means of physical activity from childhood. Among the physical exercise programs for the improvement of these variables we can highlight high-intensity interval training. However, most of these studies have been carried out on overweight or obese athletes or schoolchildren and existing protocols on high intensity intervallic training are different. The main objective of the present research is to compare two high-intensity intervallic training protocols on body composition, heart rate, blood pressure, lipid profile, blood glucose, cardiovascular fitness, strength, quality of life, physical activity, enjoyment of physical activity and accident proneness in adolescents. The present investigation will be elaborated by a randomized-control trial design, with 2 experimental groups and a control group (CG). In each experimental groups a different protocol of high-intensity interval training is applied.

It is assessed cardiovascular capacity and strength. Body composition is assessed. Heart rate and blood pressure were also recorded. Lipid profile and blood glucose were obtained by blood sampling. Quality of life, sedentary and physical activity lifestyle, enjoyment of physical activity and Psychoeducational factors determining accident process are assessed.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death today. These have been inversely correlated with physical activity and fitness in adults, children and adolescents. In this sense, certain risk factors associated with cardiovascular disease could be prevented or treated by means of physical activity from childhood. Traditionally, the benefits of physical activity on cardiovascular markers and physical fitness in children and adolescents have been described in research conducted with traditional aerobic exercise programs. Among the physical exercise programs for the improvement of these variables we can highlight high-intensity interval training. However, most of these studies have been carried out on overweight or obese athletes or schoolchildren. On the other hand, the existing protocols on high intensity intervallic training are different, there have been intensive and extensive protocols. Likewise, the investigations do not usually control the real intensity of work and it has been described that in most cases the participants do not manage to reach the described intensity, which indicates that they are not working at the level that is considered or they are working with an intensity of an extensive protocol while the duration is of an intensive protocol. In this sense, the objective of the present research is a) to know the effect of high intensity intervallic training on body composition, heart rate, blood pressure, lipid profile, glycemia, cardiovascular capacity, strength, quality of life, physical activity, enjoyment of physical activity and accident proneness in adolescents and b) to compare two high-intensity intervallic training protocols on body composition, heart rate, blood pressure, lipid profile, blood glucose, cardiovascular fitness, strength, quality of life, physical activity, enjoyment of physical activity and accident proneness in adolescents.

The present investigation will be elaborated by a randomized-control trial design, with 2 experimental groups and a control group (CG); with pre-test and post-test. Each experimental groups performance differences protocol of high-intensity interval training.

The inclusion criteria will be: a) being in Compulsory Secondary Education; b) not presenting any musculoskeletal, neurological, cardiological, metabolic, rheumatic or previous history of spinal pathologies or with previous treatment; c) be active in the sessions of Physical Education.

Primary outcome measure are cardiovascular capacity, strength of upper limbs and strength of lower limbs. These variables are tested with "Course Navette test", handgrip dynamometry and long jump test, respectively.

Secondary outcome measure are body composition and its assessed by height, weight, waist circumference, fat percentage, hydration, muscle mass, bone weight and visceral fat. The body mass index will be obtained by recording weight and height (BMI = Weight (kg) / height (cm) 2). Heart rate and blood pressure were also recorded. Lipid profile (high density lipoproteins, low density lipoproteins and triglycerides) and blood glucose were obtained by blood sampling. Quality of life are assessed through the "Kidscreen-27 questionnaire". The sedentary lifestyle as well as the level of physical activity will be evaluated through the Adolescent International Physical Activity Questionnaire (IPAQ).

The enjoyment of physical activity and a questionnaire on Psychoeducational factors determining accident proneness in adolescents were assessed.

Intensity was assessed during all sessions by means of a heart rate monitor for each adolescent.

The type of activity used to develop the training was continuous running. After the usual warm-up in physical education classes, one of the two high-intensity interval training protocols was applied. Both have the same work time but distributed in different ways and with different intensities.

The intensive high intensity intervallic training group performs 6 sets of 60 seconds of work and 60 seconds of rest. During the first two weeks we work at an intensity of 80-85% of the reserve heart rate during the work phase and 50-55% of the reserve heart rate during the rest time. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 95-95% of the reserve heart rate.

The extensive high-intensity intervallic training group performs 3 sets of 120 seconds of work and 120 seconds of rest at an intensity of 70-75% of the reserve heart rate during the work phase and an intensity of 50-55% of the reserve heart rate during the rest phase. In weeks 3 and 4 the intensity in the work phase is increased by 5%, reaching from the fifth week onwards a work intensity of 80-85% of the reserve heart rate.

The program duration is 8 weeks and the frequency of intervention is 2 sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* being in Compulsory Secondary Education
* be active in the sessions of Physical Education

Exclusion Criteria:

* presenting any musculoskeletal, neurological, cardiological, metabolic, rheumatic or previous history of spinal pathologies or with previous treatment

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change to baseline to 8 week of Cardiovascular capacity | Two times. Baseline and 8 week later
  Cardiovascular capacity is evaluated by means of the Course Navete test. A high value in this test refers to a better cardiovascular capacity.
Change to baseline to 8 week of Manual clamping force | Two times. Baseline and 8 week later
  Manual grip strength is assessed by means of dynamometry. The higher the value in this test, the greater the manual grip strength. It is recorded in kilograms.
Change to baseline to 8 week of Long jump | Two times. Baseline and 8 week later
  The long jump is recorded by means of a mobile application. A higher value in this test reflects greater strength in the lower extremities. It is recorded in centimeters.

SECONDARY OUTCOMES:
Change to baseline to 8 week of Height | Two times. Baseline and 8 week later
  The size of the subject will be measured in centimeters.
Change to baseline to 8 week of Weight | Two times. Baseline and 8 week later
  The Weight of the subject will be measured in kilograms.
Change to baseline to 8 week of Waist circumference | Two times. Baseline and 8 week later
  The waist circumference of the subject will be measured in centimeters.
Change to baseline to 8 week of Fat percentage | Two times. Baseline and 8 week later
  The percentage of fat was assessed by bioimpedance.
Change to baseline to 8 week of Hydration percentage | Two times. Baseline and 8 week later
  The hydratation was assessed by bioimpedance.
Change to baseline to 8 week of Muscle mass | Two times. Baseline and 8 week later
  The muscle mass was assessed by bioimpedance. It was register in kilograms.
Change to baseline to 8 week of Bone weight | Two times. Baseline and 8 week later
  The bone weight was assessed by bioimpedance. It was register in kilograms.
Change to baseline to 8 week of Visceral fat | Two times. Baseline and 8 week later
  The visceral fat was assessed by bioimpedance. It was register in kilograms.
Change to baseline to 8 week of Heart rate | Two times. Baseline and 8 week later
  The heart rate is taken under a blood pressure and heart rate device and the value is given in number of beats per minute.
Change to baseline to 8 week of systolic and diastolic Blood pressure | Two times. Baseline and 8 week later
  Blood pressure (systolic and diastolic) is taken under a blood pressure and heart rate measuring device and the value is given in number of millimeters of mercury.
Change to baseline to 8 week of Blood glucose | Two times. Baseline and 8 week later
  Blood glucose lipoproteins is analyzed by blood extraction.
Change to baseline to 8 week of High density lipoproteins | Two times. Baseline and 8 week later
  High-density lipoproteins is analyzed by blood extraction.
Change to baseline to 8 week of Low density lipoproteins | Two times. Baseline and 8 week later
  Low-density lipoproteins is analyzed by blood extraction.
Change to baseline to 8 week of Triglycerides | Two times. Baseline and 8 week later
  Triglycerides is analyzed by blood extraction.
Change to baseline to 8 week of Quality of life level | Two times. Baseline and 8 week later
  Quality of life was assessed through the "Kidscreen-27 questionnaire" (assess health and subjective well-being in children and adolescents). This questionnaire report a score on a scale, with 5 option (never, a little, often, very often and always). The minimum value is 0 up to 100. A higher score on this test reflects a higher quality of life level. Higher score mean a better outcome.
Change to baseline to 8 week of Sedentary and physical activity lifestyle | Two times. Baseline and 8 week later
  The sedentary lifestyle as well as the level of physical activity will be evaluated through the Adolescent International Physical Activity Questionnaire (IPAQ).
Change to baseline to 8 week of Enjoyment of physical activity | Two times. Baseline and 8 week later
  The enjoyment of physical activity was measure by a questionaire.
  This questionnaire report a score on a scale, with 5 option (strongly disagree, somewhat disagree, neutral, somewhat agree and strongly agree). The minimum value is 0 up to 100. A higher score on this test reflects a higher enjoyment. Higher score mean a better outcome.
Risk of Accident level | 8 week
  Psychoeducational factors determining accident proneness in adolescents were assessed by questionaire. A higher score on this test reflects a higher risk of an adolescent accident. The questionnaire is composed of 4 factors. Factor 1. Perceived competence (from 8 to 48 points); Factor 2. Factor 3. Competitiveness (from 4 to 24 points), Factor 4. Risk-taking (from 4 to 24 points); and Factor 5. A higher score mean a high point in the factor.

CONTACTS AND LOCATIONS:
Overall Officials: NOELIA GONZALEZ GALVEZ, PhD, Principal Investigator — UCAM
Locations (1):
- Noelia G González-Gálvez, PhD., Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Galvez N, Vaquero-Cristobal R, Macia-Andreu MJ, Garcia-Tascon M, Soler-Marin A, Gallardo-Guerrero AM. Influence of physical fitness components on personality factors and risk perception of children and adolescents: a cross-sectional study. BMJ Open. 2023 Dec 10;13(12):e071995. doi: 10.1136/bmjopen-2023-071995. PMID 38072471